CLINICAL TRIAL: NCT04408911
Title: The Effect of Lormetazepam Versus Midazolam in Critically Ill Patients on Hospital Mortality: a Retrospective Cohort Trial
Brief Title: Lormetazepam Versus Midazolam in Critically Ill Patients: a Retrospective Cohort Trial
Acronym: RetroLoveMi
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Felix Balzer, Prof. Dr. med. Dr. rer. nat. Felix Balzer, Charite University, Berlin, Germany
Other Study IDs: RetroLoveMi
Record Dates: First submitted 2020-05-22; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Midazolam: Critically ill intensive care unit patients receiving midazolam
  Interventions: Drug: Midazolam vs. Lormetazepam
- Lormetazepam: Critically ill intensive care unit patients receiving lormetazepam
  Interventions: Drug: Midazolam vs. Lormetazepam

INTERVENTIONS:
Drug: Midazolam vs. Lormetazepam — In this retrospective analysis we compared critically ill ICU patients receiving midazolam to those receiving lormetazepam.

SUMMARY:
The aim of this retrospective cohort study is to evaluate the effect of lormetazepam versus midazolam on hospital mortality, intensive care unit outcomes and sedation management.

The hypothesis is that patients receiving midazolam have a 5% higher hospital mortality in comparison to patients receiving lormetazepam.

DETAILED DESCRIPTION:
Sedation is an integral part of modern intensive care medicine and has seen a tremendous development throughout the last years. Current guideline recommendations are targeted at an awake critically ill patients (target Richmond Agitation-Sedation Scale 0/-1) as early deep sedation has been shown to negatively affect the outcome. Nevertheless, is an adequate and individualized anxiolysis still an important intervention that can be achieved via process optimization, modifications to the infrastructure of the ward and pharmacologic therapy. Bolus application of benzodiazepines is a recommended pharmacologic measure to achieve proper anxiolysis. Midazolam is currently the most commonly used benzodiazepine in European intensive care units. Midazolam accumulates after repetitive application due to its pharmacokinetic properties, which increases the likelihood for side effects and makes targeted sedation increasingly difficult. Lormetazepam is used with increasing frequency as it is eliminated independent of the patients age and has few relevant metabolites. It is therefore thought to be better suited for targeted sedation management, which in turn would be beneficial for the patients.

The aim of this retrospective cohort study is to evaluate the effect of lormetazepam versus midazolam on hospital mortality, intensive care unit outcomes and sedation management.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit patients at the Charité - Universitätsmedizin Berlin
* Age ≥ 18 years
* Intensive care unit length of stay ≥ 48 hours
* Duration of mechanical ventilation > 0 hours
* Midazolam or lormetazepam application during the ICU stay

Exclusion Criteria:

* Number of application < 2
* Midazolam and lormetazepam application during the intensive care unit stay
* Neurosurgical intensive care unit patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients at the Charité - Universitätsmedizin Berlin that received either midazolam or lormetazepam.
Sampling Method: Non-Probability Sample
Enrollment: 3314 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | On average 20 days, for each study subject measured up to study completion day 12-31-2018
  Proportion of patients that between hospital admission and hospital discharge

SECONDARY OUTCOMES:
Incidence of delirium during the intensive care unit stay | On average 7 days, for each study subject measured up to study completion day 12-31-2018
  Incidence of delirium diagnosed on the intensive care unit
Duration of delirium during the intensive care unit stay | On average 3 days, for each study subject measured up to study completion day 12-31-2018
  Duration patients had a delirium on the intensive care unit
Hospital length of stay | On average 30 days, for each study subject measured up to study completion day 12-31-2018
  Time patients spend admitted to the hospital
Intensive care unit length of stay | On average 7 days, for each study subject measured up to study completion day 12-31-2018
  Time patients spend admitted to the intensive care unit
Duration of mechanical ventilation | On average 4 days, for each study subject measured up to study completion day 12-31-2018
  Time patients are mechanically ventilated

IPD SHARING:
Plan to Share IPD: No